CLINICAL TRIAL: NCT05904522
Title: Evaluation of Histopathological Changes in the Non-lesional Skin of Stage 1A Mycosis Fungoides Patients
Brief Title: Histopathological Changes in Mycosis Fungoides
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: mf-E.84376
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Mycosis Fungoides
Keywords: mycosis fungoides; histopathology
MeSH Terms: conditions — Mycosis Fungoides | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Biopsies will be taken from lesional and non-lesional skin of the patients in the dermatology clinic and sent to laboratory for histopathologic examination. Lesional skin of the patient will be compared with the non-lesional skin of the same patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lesional skin (Experimental): lesional skin of mycosis fungoides stage 1A patients
  Interventions: Diagnostic Test: biopsy
- non-lesional skin (Experimental): non-lesional skin of mycosis fungoides stage 1A patients
  Interventions: Diagnostic Test: biopsy

INTERVENTIONS:
Diagnostic Test: biopsy — biopsy for histopathological examination

SUMMARY:
Patients with mycosis fungoides stage 1A disease have patch and plaque lesions less than %10 of body skin area. Aim of the study is to compare lesional and non-lesional skin of mycosis fungoides patients, and to decide if the systemic treatment is better or local treatment is better for them. Two biopsies for each patient were taken from lesional and non-lesional skin area.

DETAILED DESCRIPTION:
Patients with mycosis fungoides stage 1A disease have patch and plaque lesions less than %10 of body skin area. Aim of the study is to compare lesional and non-lesional skin of mycosis fungoides patients, and to decide if the systemic treatment is better or local treatment is better for them. Two biopsies for each patient were taken from lesional and non-lesional skin area.

Biopsies will be taken from lesional and non-lesional skin of the patients in the dermatology clinic and sent to laboratory for histopathologic examination.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed mycosis fungoides stage 1A patients

Exclusion Criteria:

* Mycosis fungoides patients with other stages

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
CD4+ T cells in epidermis | 6 months
  Histopathologically clonal T lymphocytes in epidermis reveal the diagnosis. If they are seen in non-lesional skin, then lesional specific local treatment is not enough for the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University Hospital, Istanbul, Turkey (Türkiye)